CLINICAL TRIAL: NCT01665898
Title: Randomized Controlled Trial Comparing Cold Biopsy Forceps Versus Cold Snare Biopsy for Colon Polyps
Brief Title: Comparing Cold Biopsy Forceps Versus Cold Snare Biopsy for Colon Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Joon Sung Kim, Instructor, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IncheonSMH; OC12OISI0067 (Other: CMCIRB)
Record Dates: First submitted 2012-08-09; First posted 2012-08-16 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Colon Polyps
Keywords: cold biopsy forceps; cold snare biopsy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cold biopsy forceps (Active Comparator): Cold biopsy forceps for removal of colon polyps
  Interventions: Procedure: Cold Biopsy forceps
- Cold Snare Biopsy (Active Comparator): Cold snare biopsy for removal of colon polyps
  Interventions: Procedure: Cold snare biopsy

INTERVENTIONS:
Procedure: Cold Biopsy forceps — removal of polyps using cold biopsy forceps
  Arms: Cold biopsy forceps
Procedure: Cold snare biopsy — Removal of colon polyps using cold snare biopsy
  Arms: Cold Snare Biopsy

SUMMARY:
Comparing the efficacy of cold biopsy forceps versus cold snare biopsy for removing colon polyps.

DETAILED DESCRIPTION:
Polyps were randomized to be treated with either CSP or CFP. After the initial polypectomy, additional EMR was performed at the polypectomy site to assess the presence of residual polyp tissue.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 40 years old and
* patients who are receiving colonoscopies and
* patients who have colon polyps

Exclusion Criteria:

* patients who have not agreed to the study
* patients with bleeding tendencies

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Comparing the complete removal rate of cold biopsy forceps versus cold snare biopsy for removing colon polyps | up to 3 years
  We will investigate the complete removal rate of colon polyps by using two different methods, cold biopsy forceps or cold snare biopsy. After removal of polyps by one of these two methods, the remnant lesion will be biopsied to study if there are any remnant tissues in order to find out the complete removal rate.

SECONDARY OUTCOMES:
Bleeding rate after removal of colon polyps by using cold biopsy forceps or cold snare biopsy | participants will be followed up for 1 month
  We will investigate bleeding rate after removal of colon polyps by these two methods. Bleeding rate will be the number of patients who showed significant bleeding after the procedure divided by the total number of patients who will receive the procedure. Significant bleeding was determined to be ongoing bleeding for more than 30 seconds after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Bo-In Lee, Principal Investigator — Incheon St.Mary's Hospital
Locations (1):
- Incheon St. Mary's Hospital, Incheon, South Korea

REFERENCES:
- [Derived] Kim JS, Lee BI, Choi H, Jun SY, Park ES, Park JM, Lee IS, Kim BW, Kim SW, Choi MG. Cold snare polypectomy versus cold forceps polypectomy for diminutive and small colorectal polyps: a randomized controlled trial. Gastrointest Endosc. 2015 Mar;81(3):741-7. doi: 10.1016/j.gie.2014.11.048. PMID 25708763